CLINICAL TRIAL: NCT03733834
Title: Comparisiom of Standard (SD) Therapy and Non-standard (NSD) Therapy in Elderly Acute Myeloid Leukemia (AML)
Brief Title: SD vs. NSD Therapy in Elderly AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University Shenzhen Hospital (Other); First Affiliated Hospital of Shenzhen University (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); First Affiliated Hospital of Guangxi Medical University (Other); Xiangya Hospital of Zhongnan University (Unknown); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Gannan Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, professor, Nanfang Hospital, Southern Medical University
Other Study IDs: Therapy in elderly AML-2018
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Standard Therapy; Non-standard Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SD therapy: SD therapy is definited as the treatment regimen must follow NCCN guildline and chemotherapy intensity could not be reduced.
- NSD therapy: Non-standard (NSD) therapy is definited as patients receiving reduced-intensity therapy or only supporting care.

SUMMARY:
It is known that treatment outcome could be positively associated with treatment intensity. However, tolerance of chemotherapy decreases in the elder, some patients could not tolerate standard (SD) therapy and even died of side effect, and overall survival (OS) might not be prolonged. Whether all elder acute myeloid leukemia (AML) patients could benefit from SD therapy, or some should receive reduced-intensity therapy or even only supporting care remains controvertal. In this multi-center study, we are going to evaluate the benefit of SD and non-SD (NSD) therapy in elder AML patients.

DETAILED DESCRIPTION:
It is known that treatment outcome could be positively associated with treatment intensity. However, tolerance of chemotherapy decreases in the elder, some patients could not tolerate standard (SD) therapy and even died of side effect, and overall survival (OS) might not be prolonged. Whether all elder acute myeloid leukemia (AML) patients could benefit from SD therapy, or some should receive reduced-intensity therapy or even only supporting care remains controvertal. SD therapy is definited as the treatment regimen must follow NCCN guildline and chemotherapy intensity could not be reduced. Non-SD (NSD) therapy is definited as patients receiving reduced-intensity therapy or only supporting care. In this multi-center study, we are going to evaluate the benefit of SD and NSD therapy in elder AML patients.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed AML exclusive of APL; Age from 60 years old to 75 years old.

Exclusion Criteria:

Any abnormality in a vital sign (e.g., organ function failure, serious infection ) Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed AML exclusive of APL with age range from 60 years old to 75 ages old. Patients are expect to live longger than 3 months.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  The time from AML diagnosis to patients death or last folloeing-up.

SECONDARY OUTCOMES:
Relapse-free survival | 2 years
  The time from AML patients obtaining CR to patients relapse or last folloeing-up.
Relapse incidence | 2 years
  Relapsed patients account for all the diagnosed AML patients.
Treatment-related mortality | 1 year
  The incidence of patients dying of treatment related complication.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China